CLINICAL TRIAL: NCT01854957
Title: MEsenchymal StEm Cells for Multiple Sclerosis (MESEMS) Phase I-II Clinical Trial With Autologous Mesenchymal Stem Cells (MSCs) for the Therapy of Multiple Sclerosis
Brief Title: MEsenchymal StEm Cells for Multiple Sclerosis
Acronym: MESEMS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Antonio Uccelli (Other)
Collaborators: Azienda Ospedaliera Universitaria Integrata Verona (Other); Ospedale San Raffaele (Other)
Responsible Party: Sponsor-Investigator, Antonio Uccelli, MD, University of Genova
Organization: University of Genova (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MESEMS; 2011-001295-19 (EudraCT Number)
Record Dates: First submitted 2013-05-08; First posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Mesenchymal stem cells
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous Mesenchymal Stem Cells (Experimental): At week 0 a single infusion of either ex-vivo expanded autologous MSC or suspension media will be administered intravenously at a dose of 1-2 x 1000000 MSC/Kg body weight. At week 24, another infusion will be performed for cross-over re-treatment: at week 24 treatments will be reversed compared to week 0
  Interventions: Biological: Autologous Mesenchymal Stem Cells
- Suspension media (Placebo Comparator): At week 0 a single infusion of either ex-vivo expanded autologous MSC or suspension media will be administered intravenously at a dose of 1-2 x 1000000 MSC/Kg body weight. At week 24, another infusion will be performed for cross-over re-treatment: at week 24 treatments will be reversed compared to week 0

INTERVENTIONS:
Biological: Autologous Mesenchymal Stem Cells — Single dose of 1-2 x 1000000 cells/Kg body weight
  Arms: Autologous Mesenchymal Stem Cells

SUMMARY:
A double-blind, randomized, cross-over phase I/II study to evaluate the safety and the efficacy of the intravenous administration of autologous Mesenchymal Stem Cells (MSC) to patients with active multiple sclerosis (MS) resistant to currently available therapies.

DETAILED DESCRIPTION:
The mechanism of action of MSC relies on their ability to modulate pathogenic immune responses and provide neuroprotection through the release of anti-apoptotic, anti-oxidant and trophic factors as demonstrated by in vitro and in vivo preclinical studies.

Patients will be randomized to receive immediate vs. delayed treatment with either a dose equal to 1-2 millions/kg of body weight of autologous MSC, or equivalent volume of suspension media at baseline. At 6 months treatments will be reversed.

The primary outcome of this study is to evaluate

* treatment's safety within one year from MSC administration by measuring the the number, time-frame and severity of adverse event and
* treatment's activity in terms of reduction in the total number of contrast-gadolinium enhancing lesions (GEL) by magnetic resonance imaging (MRI) scans.

Secondary outcomes are to gain preliminary information on the efficacy of the experimental treatment in terms of combined MRI activity and clinical efficacy (incidence of relapses and disability progression).

ELIGIBILITY:
Inclusion Criteria:

- 1. Diagnosis of MS

a. Relapsing remitting MS (RRMS) not responding to at least a year of attempted therapy with one or more of the approved therapies (beta-interferon, glatiramer acetate, natalizumab, mitoxantrone, fingolimod) as evidenced by one or more of the following: i. ≥1 clinically documented relapse in past 12 months

ii. ≥2 clinically documented relapses in last 24 months

iii. ≥1 GEL at MRI performed within the last 12 months

b. Secondary progressive MS (SPMS) not responding to at least a year of attempted therapy with one or more of the approved therapies (beta-interferon, glatiramer acetate, natalizumab, mitoxantrone, fingolimod) as evidenced by both:

i. an increase of ≥1 point of the expanded disability status scale (EDSS) (if at randomization EDSS ≤ 5.0) or 0.5 EDSS point (if at randomization EDSS ≥ 5.5) in the last 12 months

ii. ≥1 clinically documented relapse or ≥ 1 GEL at MRI within the last twelve months.

c. Primary progressive MS (PPMS) patients with all the following features:

i. an increase of ≥1 EDSS point (if at randomization EDSS ≤ 5.0) or 0.5 EDSS point (if at randomization EDSS ≥5.5), in the last twelve months

ii. ≥ 1 GEL at MRI performed within the last 12 months

iii. positive cerebrospinal fluid (CSF) (oligoclonal banding

* 2. Age 18 to 50 years
* 3. Disease duration 2 to 10 years (included)
* 4. EDSS 3.0 to 6.5

Exclusion Criteria:

* 1. RRMS not fulfilling inclusion criteria
* 2. SPMS not fulfilling inclusion criteria
* 3. PPMS not fulfilling inclusion criteria
* 4. Any active or chronic infection including infection with HIV1-2 or chronic Hepatitis B or Hepatitis C
* 5. Treatment with any immunosuppressive therapy, including natalizumab and fingolimod, within the 3 months prior to randomization
* 6. Treatment with interferon-beta or glatiramer acetate within the 30 days prior to randomization
* 7. Treatment with corticosteroids within the 30 days prior to randomization
* 8. Relapse occurred during the 60 days prior to randomization
* 9. Previous history of a malignancy other than basal cell carcinoma of the skin or carcinoma in situ that has been in remission for more than one year
* 10. Severely limited life expectancy by another co-morbid illness
* 11. History of previous diagnosis of myelodysplasia or previous hematologic disease or current clinically relevant abnormalities of white blood cell counts
* 12. Pregnancy or risk or pregnancy (this includes patients that are unwilling to practice active contraception during the duration of the study)
* 13. eGFR < 60 mL/min/1.73m2 or known renal failure or inability to undergo MRI examination.
* 14. Inability to give written informed consent in accordance with research ethics board guidelines

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Safety | 24 weeks from the first infusion
  Incidence and severity of adverse events in MSC treatment group compared to placebo group.
efficacy | 24 weeks from the first infusion
  total number of contrast-enhancing lesions (GEL) at MRI scan

SECONDARY OUTCOMES:
Efficacy | 48 weeks from the first infusion
  Number of GEL counted over week 28, 36 and 48 compared with the number of GEL counted over 4, 12 and 24 weeks.
Efficacy | 24 weeks form the first infusion
  Combined unique MRI activity (number of new or enlarging T2, or enhancing or re-enhancing lesions), volume of GEL and volume of black holes (BH) over 4, 12, 24 weeks compared between treatment groups.
Efficacy | 48 weeks from the first infusion
  Combined unique MRI activity, volume of GEL and volume of BH over week 28, 36 and 48 compared with the same outcomes over 4, 12 and 24 weeks.
Efficacy | 48 weeks from the first infusion
  Number of relapses in MSC treatment group vs. placebo group in the first 24 weeks and after cross-over re-treatment in the two groups.
Efficacy | 48 weeks from the first infusion
  Time to sustained progression of disability and proportion of progression-free patients compared between treatment groups during the first 24 weeks and after cross-over

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Comi, MD, Principal Investigator — Ospedale San Raffaele; Bruno Bonetti, MD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata di Verona
Locations (1):
- University of Genova, Genova, Genova, Italy

REFERENCES:
- [Derived] Thebault S, Reaume M, Marrie RA, Marriott JJ, Furlan R, Laroni A, Booth RA, Uccelli A, Freedman MS. High or increasing serum NfL is predictive of impending multiple sclerosis relapses. Mult Scler Relat Disord. 2022 Mar;59:103535. doi: 10.1016/j.msard.2022.103535. Epub 2022 Jan 19. PMID 35078125
- [Derived] Uccelli A, Laroni A, Brundin L, Clanet M, Fernandez O, Nabavi SM, Muraro PA, Oliveri RS, Radue EW, Sellner J, Soelberg Sorensen P, Sormani MP, Wuerfel JT, Battaglia MA, Freedman MS; MESEMS study group. MEsenchymal StEm cells for Multiple Sclerosis (MESEMS): a randomized, double blind, cross-over phase I/II clinical trial with autologous mesenchymal stem cells for the therapy of multiple sclerosis. Trials. 2019 May 9;20(1):263. doi: 10.1186/s13063-019-3346-z. PMID 31072380